CLINICAL TRIAL: NCT01842724
Title: Motec Versus Remotion Total Wrist Arthroplasty - A Prospective Randomized Study.
Brief Title: Motec Versus Remotion Total Wrist Arthroplasty - A Prospective Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trygve Holm Glad, MD, Oslo University Hospital
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 2013/149
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Non-rheumatoid Wrist Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motec total wrist arthroplasty (Active Comparator)
  Interventions: Procedure: Motec total wrist arthroplasty
- Remotion total wrist arthroplasty (Active Comparator)
  Interventions: Procedure: Remotion total wrist arthroplasty

INTERVENTIONS:
Procedure: Motec total wrist arthroplasty
  Arms: Motec total wrist arthroplasty
Procedure: Remotion total wrist arthroplasty
  Arms: Remotion total wrist arthroplasty

SUMMARY:
The purpose of this study is to determine the difference in the results between Motec and Remotion wrist arthroplasty in the treatment of non-rheumatoid wrist arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful non-rheumatoid wrist arthritis (posttraumatic arthritis and late stage Kienboeck's disease)
* Age 18-70 years
* ASA class 1-3

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2034-11 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
PRWHE (Patient rated Wrist and Hand Evaluation score) | 24 months postop
  PRWHE is a wrist specific patient assessed questionnaire, measuring pain, wrist specific function and general function

SECONDARY OUTCOMES:
Wrist movement | 24 months postop
  Overall degree of flexion, extension, radial and ulnar deviation
Grip Strength | 24 months postop
Pain in affected wrist | 24 months postop
  Visual analogue scale
Quick-DASH | 24 months postop
  "Disabilities of the Arm, Shoulder and Hand" questionnaire
intraoperative complications | intraoperative
Postoperative complications | 24 months postop
Implant loosening | 24 months postop
  Implant loosening seen on x-ray
Implant migration | 24 months postop
  Implant migration seen on model-based roentgen stereophotogrammetric analysis (RSA), as a possible precursor of later implant loosening
Periprosthetic bone mineral density | 24 months postop
  BMD measured with DEXA (dual-energy x-ray absorptiometry)
Reoperations | 24 months postop
  Reoperations of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Trygve Holm Glad, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway